CLINICAL TRIAL: NCT05527990
Title: A Study of Next-generation Pulse Oximeters to Support the Integrated Management of Childhood Illnesses in Primary Care Settings. A Mixed Methods Type 2 Effectiveness-implementation Study Measuring the Performance and Feasibility, of Multimodal Pulse Oximeter Devices by Primary Care Providers
Brief Title: TIMCIs: A Hybrid Type 2 Study of Next-generation Pulse Oximeters
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: PATH (Other)
Collaborators: UNITAID (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: RES-00317
Record Dates: First submitted 2022-08-30; First posted 2022-09-06 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Focus of Study: Accurate Clinical Measurement and Diagnosis
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Multimodal PO — Mixed methods diagnostic accuracy and implementation of multimodal PO

SUMMARY:
This study aims to provide evidence on next-generation clinical measurement tools through a mixed methods diagnostic accuracy and implementation study in Kenya, Senegal, Tanzania, and Uttar Pradesh, India.

DETAILED DESCRIPTION:
Performance and feasibility of photoplethysmograph (PPG)-derived clinical measurement tools (medical device and smartphone-based screening technologies) by primary care providers will be assessed using a type 2 hybrid design to conduct a mixed methods diagnostic accuracy and implementation study.

The diagnostic accuracy study will consist of 3 components to achieve the primary and secondary objectives: 1) a usability assessment of observed user-product interactions and a system usability score, 2) measurement of multimodal PO device performance through comparison against a reference standard, and 3) caregiver/provider acceptability through semi-structured interviews.

The observational implementation (OI) study consists of 3 components to achieve the primary and secondary objectives: 1) a human-centered design workshop, 2) an observational study to evaluate the feasibility of implementing an approved multimodal PO device in clinical care, and 3) semi-structured in-depth interviews to assess provider and caregiver acceptability and adaptation.

The interventions for this study are PPG-derived clinical measurement tools that measure oxygen saturation (SpO2), pulse rate, respiratory rate, and/or temperature. The interventions will also be compared to a reference standard for the different clinical measurements

ELIGIBILITY:
Inclusion Criteria:

* Children 0 - 59 months for whom caregivers provide consent to participate in the research study, following completion of clinical consultation
* Consulting for a respiratory illness, or reported to have a respiratory illness when attending for a routine visit as an outpatient (e.g., vaccination, growth, or chronic disease monitoring)

Exclusion Criteria:

* Children in the immediate post-natal period or first day of life
* Attending for a consultation related to trauma only (including new and follow-up presentations for burns, injuries, wounds)
* Admitted within an inpatient part of the facility (including neonates delivered at the facility admitted with their mother)
* Children who are critically ill, requiring emergency treatment, or received a recommendation of immediate referral during clinical consultation

Max Age: 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 0 - 59 months consulting for or reported to have a respiratory illness.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2022-03-20 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy: Performance of clinical measurement tools | 19 weeks
  To determine the performance of PPG-derived clinical measurement tools (medical device and smartphone-based screening technologies) compared to an accepted reference standard, among children 0-59 months seeking care at the primary care level.
Observational implementation: multimodal (MM) operational feasibility | 16 weeks
  To evaluate the operational feasibility of implementing an approved next generation pulse oximeter at the primary care level.

SECONDARY OUTCOMES:
DA: MM Usability | 2 weeks
  To measure the usability of multimodal PO devices, measuring pulse oximetry and respiratory rate in addition to other relevant clinical measurements, by healthcare providers at the primary care level.
DA: MM Acceptability | 21 weeks
  To assess the acceptability of multimodal PO devices among healthcare providers and caregivers at the primary care level.
DA: Data repository | 19 weeks
  To create an open-source data repository for future research on PPG-derived clinical measurement tools for children.
OI: MM/clinical measurement system requirements | 16 weeks
  To explore future multimodal PO device and smartphone based clinical measurement product concepts and prototypes to further define the user and health system requirements for potential device integration within integrated management of childhood illness (IMCI) care practices, among country stakeholders and healthcare providers.
OI: MM co-design | 1 week
  To co-design integration of an approved multimodal PO device within existing IMCI practices, mapping current and future state workflows, prioritizing outcomes, and determining training needs.

CONTACTS AND LOCATIONS:
Locations (2):
- Kenya (2):
  - Mathare North Health Center, Nairobi
  - Ngiri Health Center, Nairobi

IPD SHARING:
Plan to Share IPD: No